CLINICAL TRIAL: NCT04518384
Title: Risk Factors Associated With Anastomotic Leak and Perioperative Mortality in Elderly Patients Undergoing Colorectal Surgery.
Brief Title: Risk Factors Associated With Anastomotic Leak and Perioperative Mortality in Elderly
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, ilan schrier, Dr. Ilan Schrier, Rabin Medical Center
Other Study IDs: 0441-17-RMC
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colon or rectum resection — surgical procedure to resect the colon or rectum

SUMMARY:
This is a retrospective cohort study of all consecutive patients who underwent colon or rectal resection, between the years 2012-2017 at Rabin Medical Center, a tertiary referral center in Israel. Data were obtained from patients' electronic medical files. The study was approved by the Institutional Review Board (IRB) of Rabin Medical Center (RMC). The study met the guidelines outlined in the Declaration of Helsinki. Due to the minimal risk nature of this study, the need for informed consent was waived by the IRB.

Patient population:

All patients aged 70 years and above who underwent large bowel resection were included in the analysis. Inclusion criteria were: age ≥70; all patients undergoing any colonic or rectal resection for benign or malignant etiologies in an open or minimally-invasive approach Exclusion criteria were: age<70; colon resection without anastomoses; re-operations during the same admission .

Data retrieved included demographic data (age, gender, Charlson comorbidity score, place of residency, functional capacity, BMI), surgical data (indication for surgery, elective vs urgent surgery, surgical approach, length of surgery, peri-operative morbidity and mortality.All surgeries were performed by at least one senior surgeon. The surgical approach (laparoscopic or laparotomy) was at the senior surgeon's discretion and deemed most appropriate for the patient's problem, physiological status and underlying illnesses. The extent of the resection was according to oncological guidelines when relevant

Endpoints:

Primary endpoint was the occurrence of postoperative anastomotic leak. Secondary end-point was postoperative mortality Statistical Analysis The statistical analysis for this paper was generated using SAS Software. Continuous variables were presented by Mean±Std, Categorical variables were presented by (N, %). T-Test was used to compare the value of continuous variables between study groups and Fisher's exact test (for two groups) or Chi-square (for more than two groups) were used to compare the value of categorical variables between study groups. Two-sided p values less than .05 were considered statistically significant

DETAILED DESCRIPTION:
This is a retrospective cohort study of all consecutive patients who underwent colon or rectal resection, between the years 2012-2017 at Rabin Medical Center, a tertiary referral center in Israel. Data were obtained from patients' electronic medical files. The study was approved by the Institutional Review Board (IRB) of Rabin Medical Center (RMC). The study met the guidelines outlined in the Declaration of Helsinki. Due to the minimal risk nature of this study, the need for informed consent was waived by the IRB.

Patient population:

All patients aged 70 years and above who underwent large bowel resection were included in the analysis. Inclusion criteria were: age ≥70; all patients undergoing any colonic or rectal resection for benign or malignant etiologies in an open or minimally-invasive approach Exclusion criteria were: age<70; colon resection without anastomoses; re-operations during the same admission .

Data retrieved included demographic data (age, gender, Charlson comorbidity score, place of residency, functional capacity, BMI), surgical data (indication for surgery, elective vs urgent surgery, surgical approach, length of surgery, peri-operative morbidity and mortality.All surgeries were performed by at least one senior surgeon. The surgical approach (laparoscopic or laparotomy) was at the senior surgeon's discretion and deemed most appropriate for the patient's problem, physiological status and underlying illnesses. The extent of the resection was according to oncological guidelines when relevant.

Endpoints:

Primary endpoint was the occurrence of postoperative anastomotic leak. Secondary end-point was postoperative mortality Statistical Analysis The statistical analysis for this paper was generated using SAS Software. Continuous variables were presented by Mean±Std, Categorical variables were presented by (N, %). T-Test was used to compare the value of continuous variables between study groups and Fisher's exact test (for two groups) or Chi-square (for more than two groups) were used to compare the value of categorical variables between study groups. Two-sided p values less than .05 were considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

age ≥70; all patients undergoing any colonic or rectal resection for benign or malignant etiologies in an open or minimally-invasive approach -

Exclusion Criteria:

- age<70; colon resection without anastomoses; re-operations during the same admission .

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: age ≥70; all patients undergoing any colonic or rectal resection for benign or malignant etiologies in an open or minimally-invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2017-08-06 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
anastamotic leak | 30 days

SECONDARY OUTCOMES:
mortality | untill 8.2020

CONTACTS AND LOCATIONS:
Overall Officials: ilan schrier, MD, Principal Investigator — TAU
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No